CLINICAL TRIAL: NCT01172483
Title: Effectiveness of Community-Based Physiotherapy in Chronic Disorders Versus General Practice in Primary Care. Multicenter Randomized Control Trial
Brief Title: Effectiveness of Community-Based Physiotherapy Versus General Practice
Acronym: ECACOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Collaborators: Andaluz Health Service (Other Government)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, PhD, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 04-2009
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2013-01

CONDITIONS: Chronic Disorders
Keywords: primary care; physical and aquatic exercises; promotion physical activity; chronic disorders
MeSH Terms: conditions — Chronic Disease | interventions — Primary Health Care; Educational Status

STUDY DESIGN:
Intervention Model Description: Education & exercise
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- multimodal community program (Experimental): multimodal community program of exercise and education
  Interventions: Other: Multimodal community program
- active control (Active Comparator): general practice in primary care and education of chronic disorders
  Interventions: Procedure: general practice in primary care and education

INTERVENTIONS:
Procedure: general practice in primary care and education — education of chronic disorders in PC
  Arms: active control
Other: Multimodal community program — The intervention was an 8-week programme of MMPP combined with DWR, delivered by physiotherapists in groups of 8 to 10 participants. One-hour sessions were conducted 3 times per week, consisting of DWR and an individualised MMPP of therapeutic exercises combined with education based on cognitive-behavioural principles. Each session was comprised of 30 minutes of land-based exercise followed by 20 minutes of DWR, with an additional 10 minutes of warm-up and cool-down time. Deep water running stimulates running using a flotation device in water levels over head height. During the first two weeks of the intervention, participants undertook a low-intensity adaptation interval to learn proper exercise technique. For the remaining six weeks, participants were instructed to maintain a constant speed to achieve the prescribed HRAT. If experiencing pain while exercising, participants were asked to temporarily reduce intensity and return to target HR as capable.
  Other Names: 8-week programme of MultiModal Physiotherapy Program combined with Deep water running exercise
  Arms: multimodal community program

SUMMARY:
Summary: (Objectives and methodology of the project) AIM: To evaluate the clinical effectiveness of Community physiotherapy intervention on chronic diseases (heart disease, chronic obstructive pulmonary disease, back pain, mechanical neck pain, fibromyalgia, osteoarthritis lower limbs, neurological and cancer survivors) and a group of healthy patients cardiovascular risk factors. DESIGN: Randomized, controlled, prospective study. SUBJECTS OF STUDY: Patients with chronic disease go to the Local Sports Torremolinos Center INTERVENTION: Establishment of a control group that give you some advice education care (brief advice) and a group common experimental multimodal program of 12 weeks therapeutic exercise with health education (brief advice). It will follow up complete with ratings pre and post intervention to both groups and follow up at 6 and 12 months for long-term effect through specific questionnaires for each subgroup chronic disease and pain score (visual scale analog), quality of life (EuroQol-5D) and state health general (Short-Form 12, SF-12) VARIABLES: The intervention physical therapy Community. Result: Specific questionnaires for each subgroup, pain (Visual analogue scale), quality of life (EuroQoL) and general health status (SF-12). DATA ANALYSIS: descriptive statistics, measuring central tendency and dispersion of the variables study. Inferential statistics will be made between intervention of key variables and outcome (Chi square, Student t, ANOVA, Mann-Whitney, Wilcoxon, by type and normal variables). Likewise, establish measures of effect size in main outcome variables, by reduction relative risk, absolute risk and odds ratio with their respective confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria will be severe cuts of the disease based on functionality and not the dysfunction indicates the severity level higher 20% of the specific questionnaire for each subgroup

Exclusion Criteria:

* Common exclusion criteria for subgroups:

"Rejection of the patient to take part in the survey

* Processes of infectious, neoplastic, metastasis, osteoporosis, inflammatory arthritis or fractures "Cognitive impairment of any etiology Presence of unstable angina, arrhythmia, unstable, failure of cardiac valvular "Severe hypertension (systolic> 200 or diastolic> 120)
* Depressed systolic function at rest (EF less than 50%)
* Evidence of exercise-induced ischemia
* Evidence of exercise-induced arrhythmias.
* Stenotic coronary lesions greater than 50%. Exercise intolerance, or physical activity any cause.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2009-12; Primary Completion 2013-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
International Physical activity Questionnaire | IPAQ
  CRAIG, C. L., A. L. MARSHALL, M. SJÖSTRÖM, A. E. BAUMAN, M. L. BOOTH, B. E. AINSWORTH, M. PRATT, U. EKELUND, A. YNGVE, J. F. SALLIS, and P. OJA. International Physical Activity Questionnaire: 12-Country Reliability and Validity. Med. Sci. Sports Exerc., Vol. 35, No. 8, pp. 1381-1395, 2003.

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire | FIQ
Minnesota living with heart failure questionnaire | MLHFQ
Saint George questionnaire | SGQ
Barthel Index | BI
WOMAC questionnaire | WOMAC
Neck Disability Index | NDI
Roland Morris Questionnaire | RMQ
PIPER CANCER-RELATED FATIGUE | Piper Fatigue Scale-Revised (PFS-R)
  The Piper Fatigue Scale-Revised (PFS-R). This 22-item self-report questionnaire asks respondents to rate their fatigue from 0 ("no fatigue") to 10 ("extreme") in 4 different domains: behavioral/severity, affective meaning, sensory and cognitive/mood.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio I Cuesta-Vargas, PhD, Principal Investigator — University of Malaga; Josefa Sanpedro, PhD, Study Director — Andalusian Health Service
Locations (1):
- Patronato Municipal de deportes de Torremolinos, Torremolinos, Malaga, Spain

REFERENCES:
- [Derived] Martin-Valero R, Cuesta-Vargas AI, Labajos-Manzanares MT. Effectiveness of the physical activity promotion programme on the quality of life and the cardiopulmonary function for inactive people: randomized controlled trial. BMC Public Health. 2013 Feb 12;13:127. doi: 10.1186/1471-2458-13-127. PMID 23399032